CLINICAL TRIAL: NCT05032651
Title: Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH)
Brief Title: Use of a Novel Artificial Intelligence Assisted Platform to Assess Optimal Dosing and Treatment Strategy of Erythropoiesis-stimulating Agents (ESA) in Hemodialysis Patients
Acronym: AI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: National Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: KMUHIRB-F(I)-20210040
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-06

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: End Stage Renal Disease; Erythropoiesis stimulating agent; Artificial intelligence assisted platform
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Randomization period All eligible subjects will be randomized 1:1 by their age, gender, and HD vintage into control arm and intervention arm. After randomization, the study subject will enter the study after the nearest Hb measurement coming.
  Study period
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A-AI (model) Arm Description: (Experimental): Artificial intelligence assisted platform supported system for the clinical physicians to prescribe ESA dose to maintain hemoglobin at the treatment target of 10 g/dl to 12 g/dl.
  Interventions: Device: novel artificial intelligence assisted platform
- GROUP B-AI (model) Arm Description: (Experimental): ESA dose prescribed by clinical physicians as regular care to maintain hemoglobin at the treatment target of 10 g/dl to 12 g/dl.
  Interventions: Device: novel artificial intelligence assisted platform

INTERVENTIONS:
Device: novel artificial intelligence assisted platform — Use of a novel artificial intelligence assisted platform

SUMMARY:
It has been known well for a long time that End stage renal disease (ESRD) patients usually need ESA to maintain their hemoglobin (Hb) to improve both mortality as well as quality of life. Later, several large-scale RCTs showing normalization of Hb in this population increased the risk of thromboembolic event, which leaded current guidelines to recommend the therapeutic goal for anemia in ESRD should be within a range (usually between 10-12 gm/dl) rather than above or below a certain level (or value). In addition to ESA dose, many factors contribute to the severity of anemia in this population, such as iron status, chronic blood loss, adequacy of dialysis, chronic inflammation, renal wasting, et al. To put all these factors together, maintaining the Hb levels within the target level is a challenge to physician. It was reported that only one third of Hb within the target at any given time. Our data showed, for those under maintenance hemodialysis and without any blood transfusion in observation period, near two third of patients' Hb level were within the target range.

DETAILED DESCRIPTION:
For better anemia management, NKF-K/DOQI developed and published guidelines using protocol or algorithm for EPO prescription.6 Recently, artificial intelligence (AI) has been widely applied to medicine in the field of reducing human error, robotic surgical system and decision- making aid. Since then, there were several studies working on decision making programs to set up model of predicting the ESA dose needed for target Hb level. Artificial neural network (ANN) model is most commonly used for ESA dose-response prediction. However, the effectiveness of these kinds of AI is not confirmed clinically and the result not satisfactory. In other words, it is still inconclusive whether contemporary AI has any role in decision making aid when prescribing ESA dose for dialysis patient, a typical trial and error which AI supposed should be very helpful with.

Based on the mentioned above, we are going to conduct this clinical try to test the hypothesis that AI is not inferior to physician in prescribing ESA dose for hemodialysis patients to maintain hemoglobin(Hb) level to meet the target

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent
2. Age older than 20 year old.
3. End stage renal disease under regular hemodialysis with three times per week and duration of each session at least 4 hours
4. Having at least consecutive 6 months data of both Hb and biochemical study during dialysis before enrollment and at least one Hb level within the range of 11-12 g/dl
5. Having at least one prescription of ESA supplement to keep Hb within the range of 10-12 g/dl in the past 6 months before the enrollment
6. Having received ESA of the same brand at least 6 months before the enrollment

Exclusion Criteria:

1. Ever receiving blood transfusion in the past 12 months
2. Active bleeding with blood loss more than 250cc in 3 months before the enrollment
3. Active infection or malignancy
4. Study subject can not follow with the study protocol

End of Study

The eligible subject will not be allowed to continue the study once informed consent is withdrawn or event happening meets the following criteria:

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
hemoglobin (Hb) levels | 6 monthes
  Maintain hemoglobin at the treatment target of 10 g/dl to 12 g/dl.

SECONDARY OUTCOMES:
the target range (10-12gm/dl) | 6 monthes
  The Proportion of Participants with haemoglobin within the target range (10-12gm/dl)
The Proportion of Participants Who Received a Whole Blood or Red Blood Cell Transfusion | 6 monthes
  The Proportion of Participants Who Received a Whole Blood or Red Blood Cell Transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hsun Wu, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided